CLINICAL TRIAL: NCT03382522
Title: Prognostic Value of SPECT-CT Quantitative Indices for the Response Assessment of Bone Metastatic Prostate Carcinoma
Acronym: INTEVOPROSTATE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: INTEVO-PROSTATE (29BRC17.0189)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: bone scintigraphy; quantification; prostate cancer; prognosis
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prognostic interest of bone scintigraphy in bone metastatic prostate carcinoma (BMPC) has been shown. Recent technological advances allow to perform quantitative bone SPECT-CT in routine practice. The aim of this study is to assess the prognostic interest of quantitative bone SPECT-CT in BMPC.

DETAILED DESCRIPTION:
Prostate adenocarcinoma is one of the most common cancer in men, and bone its most frequent distant metastasis location. 5-year survival has greatly increased these last two decades, with wide differences between countries. Nevertheless, the prognosis of castrate-resistant bone metastatic prostate cancer (BMPC) remains poor.

PCWG (Prostate Cancer Working Group) 2 has proposed in 2007 criteria to evaluate response to treatment for prostate cancer. There are based on composite data, including clinical signs (such as general condition and bone pain), Prostatic Specific Antigen (PSA) variation, CT scan (RECIST criteria) and bone scan. The scintigraphic part is based on whole body planar acquisition, and on the assessment of new uptakes. These bone scan criteria are simplistic, because only a visual analysis is possible, without consideration of changes in intensity. Moreover, these criteria consider the bone scan as a planar imaging, and it has been shown that Single Photon Emission Computed Tomography (SPECT) improved sensitivity, specificity, positive and negative predictive values in oncologic context. Finally, "PCWG2 (Prostate Cancer Working Group 2) recognizes that there are no validated criteria for response on radionuclide bone scan".

To reflect bone metastasis burden, a quantitative analysis method for bone scintigraphy, the Bone Scan Index (BSI), had been tested. BSI is based on the uptake of whole body planar imaging. While baseline BSI seemed to offer a poor correlation with overall survival (OS), on-treatment changes in BSI appeared to be a decent response marker. But a volumetric quantitative biomarker may improve the accuracy of this assessment.

The recent development of a new SPECT quantification tool (xSPECT Quant® tool, Siemens) could offer good performances on therapeutic assessment. The objective of this study is to assess the interest of this new quantitative volumetric method in bone scan response evaluation of BMPC.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent a bone SPECT-CT (Symbia INTEVO T6) between april 2014 and april 2017, with bone metastatic prostate cancer.

No opposition of the patient to participate in the study.

Exclusion Criteria:

Opposition of the patient. Age<18 y/o

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone metastatic prostate cancer Quantitative bone SPECT-CT available
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Prognostic interest of the quantitative therapeutic evaluation with bone SPECT-CT in bone metastatic prostate cancer | 3 years
  Assessment of prognostic quantitative SPECT-CT parameters

SECONDARY OUTCOMES:
Correlation between baseline quantitative bone SPECT-CT values and baseline PSA | 3 years
  Assessment of correlation between baseline PSA and baseline quantitative SPECT-CT parameters (SUVmax (max Standardized Uptake Value) of the target lesions, SUVpeak of the highest uptake lesion, Neoplastic Osteoblastic Metabolism Volume, Total Lesion Osteoblastic Metabolism) (Spearman coefficient)
Correlation between baseline quantitative bone SPECT-CT values and survival | 3 years
  Assessment of correlation between survival (Progression Free Survival, Overall Survival, Disease Specific Survival) and baseline quantitative SPECT-CT parameters (SUVmax of the target lesions, SUVpeak of the highest uptake lesion, Neoplastic Osteoblastic Metabolism Volume, Total Lesion Osteoblastic Metabolism)
Correlation between variations of quantitative bone SPECT-CT values and variations of PSA | 3 years
  Assessment of correlation between variations of PSA and variations of quantitative SPECT-CT parameters (SUVmax of the target lesions, SUVpeak of the highest uptake lesion, Neoplastic Osteoblastic Metabolism Volume, Total Lesion Osteoblastic Metabolism) (Spearman coefficient)
Correlation between variations of quantitative bone SPECT-CT values and survival | 3 years
  Assessment of correlation between survival (Progression Free Survival, Overall Survival, Disease Specific Survival) and variations of quantitative SPECT-CT parameters (SUVmax of the target lesions, SUVpeak of the highest uptake lesion, Neoplastic Osteoblastic Metabolism Volume, Total Lesion Osteoblastic Metabolism)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France